CLINICAL TRIAL: NCT01708109
Title: Optimal Handling of Common Bile Duct Calculus, a Prospective Randomized Study
Brief Title: Optimal Handling of Common Bile Duct Calculus, a Prospective Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruting patients to the study
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); Danderyd Hospital (Other); Sodertalje Hospital (Other); Mora Hospital (Unknown); Regional Hopspital Ryhov, Jönköping (Unknown); University Hospital, Linkoeping (Other); Vrinnevi Hospital, Norrköping (Unknown); Sundsvalls Hospital (Unknown)
Responsible Party: Principal Investigator, Anders Thorell, Ass. Prof., Karolinska Institutet
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/873-31/3
Record Dates: First submitted 2012-10-09; First posted 2012-10-16 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Cholelithiasis
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biliary calculus remain (Experimental): biliary calculus, less than or equal to 6 mm, remains
  Interventions: Other: no measures taken to clear bile ductus
- Biliary calculus removed (Experimental): biliary calculus, less than or equal to 6 mm, removed
  Interventions: Procedure: clearance of bile ductus

INTERVENTIONS:
Other: no measures taken to clear bile ductus — biliary calculus remain
  Arms: Biliary calculus remain
Procedure: clearance of bile ductus — biliary calculus removed at surgery
  Arms: Biliary calculus removed

SUMMARY:
The purpose is to study natural process of gallstones in common bile duct, stones less than or equal to 6 mm. And if the gallstones give any complications under 1 year follow up. The second outcome is to study side-effects of gallstones removed with surgery.

ELIGIBILITY:
Inclusion Criteria:

* cholecystectomy

Exclusion Criteria:

* Ongoing icterus or pancreatitis
* History of anamneses pancreatitis/icterus
* Allergy against x-ray contrast
* Stones more than 6 mm in ductus
* No passage of contrast to duodenum
* malignant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-11-27 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Natural process of biliary calculus left after cholecystectomy | 12 month post op
  Calculus in common bile duct less than or equal to 6 mm found during cholecystectomy, randomized to either remain or removed

SECONDARY OUTCOMES:
Complications biliary calculus | 12 month post op
  Calculus in common bile duct less than or equal to 6 mm found during cholecystectomy, randomized to either remain or removed

CONTACTS AND LOCATIONS:
Overall Officials: Anders Thorell, Assoc Prof, Principal Investigator — Karolinska Institutet
Locations (9):
- Sweden (9):
  - Regional Hospital Ryhov, Jönköping
  - Linköping University Hospital, Linköping
  - Mora Hospital, Mora
  - Vrinnevi Hospital Norrköping, Norrköping
  - Södertälje Hospital, Södertälje
  - Ersta sjukhus, Stockholm
  - Karolinska University Hospital, Stockholm
  - Danderyds Hospital, Stockholm
  - Sundsvalls Hospital, Sundsvall